CLINICAL TRIAL: NCT03950362
Title: Bladder PREserVation by RadioTherapy and Immunotherapy in BCG Unresponsive Non-muscle Invasive Bladder Cancer
Acronym: PREVERT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: prevert-IPC 2018-046
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Non-muscle-invasive Bladder Cancer
Keywords: non-muscle-invasive bladder cancer; radiotherapy; immunotherapy; quality of life
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — avelumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy associated to immunotherapy (Experimental): * Radiotherapy: 60-66 Gy in 30-33 Fractions (2 Gy/fractions) given to the whole bladder
  * Concomitant administration of Avelumab 10mg/kg Infuse IV over 30-minutes: 1 cycle 5 days before External Beam RadioTherapy, then every 21 days x 8 cycles (6 months)
  Interventions: Drug: Avelumab; Device: Radiotherapy

INTERVENTIONS:
Drug: Avelumab — Administration of Avelumab 10mg/kg Infuse IV over 30-minutes: 1 cycle 5 days before External Beam RadioTherapy, then every 21 days x 8 cycles (6 months)
Device: Radiotherapy — 60-66 Gy in 30-33 Fractions (2 Gy/fractions) given to the whole bladder

SUMMARY:
About two-thirds of newly diagnosed cases of bladder cancer are non-muscle-invasive bladder cancer (NMIBC). It is advocated that patients with high-risk NMIBC receive an adjuvant course of intravesical Bacille Calmette-Guerin (BCG) as first-line treatment. However, a substantial proportion of patients will 'fail' BCG. Radical cystectomy remains the treatment of choice for NMIBC who have failed intravesical therapy, but there are situations when surgery is not feasible due to competing co-morbidities or a patient's desire for bladder preservation. For these patients, the potential options available are limited.

In MIBC, radiotherapy (RT) in association with chemotherapy, has been shown to produce 10-year overall survival rates comparable to those of radical cystectomy in selected cases. At the opposite, results from trials assessing radiotherapy with or without chemotherapy in patients with NMIBC are less documented and discordant.

Immunotherapy with immune-checkpoint blockade therapies is increasing as an option and has shown very promising results for several cancers, including bladder carcinoma.

An established body of published work has shown that radiation enhances many of the steps needed for the generation of antigen-specific immune responses, including inflammatory tumor-cell death, dendritic cell activation, and antigen cross-presentation. Several groups have reported improved local control when checkpoint blockade immunotherapy is added to radiation in different tumor types. On the one hand, radiotherapy might stimulate the induction of local endogenous immune responses by anti-PD-1 treatment. On the other hand, active immune stimulation by anti-PD-1 treatment within the tumor microenvironment might maximize radiation-induced antitumor immunity.

Combination immunoradiotherapy using PD-1/PD-L1 signaling blockade could therefore offer an interesting strategy in bladder tumors, especially as an optional bladder preservation treatment for BCG unresponsive NMIBC.

The originality of the therapeutic strategy is the use of radiation (local treatment) combined with checkpoint blockade immunotherapy (systemic treatment). Radiotherapy might increase response rates by creating a more permissive tumor microenvironment through increasing PD-L1 expression on tumor cells and stimulating the accumulation and activation of CD8+ T cells.

Avelumab seems to have a specific cytotoxic activity suggesting its interest in local control of the disease, especially in association with radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* ECOG performance status ≤2.
* Patients having provided written informed consent prior to any study-related procedures.
* Life expectancy ≥ 12 months.
* High risk NMIBC (high grade, T1, or CIS) histologically confirmed by a systematic 2nd look complete re-TURBT.
* BCG unresponsive NMIBC defined as persistent high-grade disease at 6 months despite adequate BCG treatment (BCG refractory) or recurrence of high-grade disease within 6 months of the last BCG exposure (BCG relapsing disease).
* Inclusion within 9 months after last BCG exposure.
* Patient unfit for radical cystectomy because of age, comorbidities, or patient's refusal.
* No sign of pelvic involvement or distant metastasis on CT scan.
* Haematological and biological parameters allowing pelvic radiotherapy and anti-PDL1 administration:

  * White blood cell count ≥4000/mm3
  * Platelet count ≥100000 cells/mm3
  * Haemoglobin level ≥9 g/dL or corrected after transfusion
  * Glomerular filtration rate ≥25 mL/min.
  * Adequate hepatic function: AST (SGOT) and ALT (SGPT) ≤2.5 x ULN, or ≤3.5 x ULN in the case of concurrent disease with known etiology and for which a corrective treatment is possible.
* Patients of childbearing potential: use of a medically acceptable method of contraception during the study and for 120 days after the last study treatment.
* Patients affiliated to the social security scheme.
* Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study procedures indicated in the protocol.

Exclusion Criteria:

* Stage ≥pT2 tumors.
* Low grade recurrence / Ta recurrence after BCG therapy.
* Recurrence > 1 year after last BCG instillation.
* Prior pelvic irradiation.
* Histology other than urothelial or squamous cell carcinomas (e.g., adenocarcinomas, micropapillary, sarcomas, or small cell histological types).
* History of neoplastic disease, during the 3 years before registration, except completely resected cutaneous basal-cell carcinomas, carcinoma in-situ or localized prostate cancer without biochemical recurrence following definitive treatment.
* Prior treatment with CD137 agonists or immune checkpoint inhibitors, including anticytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4), anti-programmed death-1 receptor (anti-PD-1), and anti-programmed death-ligand 1 (anti-PD-L1) therapeutic antibodies.
* Contraindications for pelvic radiotherapy (e.g., inflammatory bowel disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
High-risk recurrence-free survival at 1 year | 1 year
  Delay between date of inclusion and reappearance of high-risk disease (high grade, T1, or CIS) at cystoscopy

IPD SHARING:
Plan to Share IPD: No